CLINICAL TRIAL: NCT00194896
Title: Rosiglitazone Intervention Study in Patients With Type 1.5 Diabetes
Brief Title: Preferred Treatment of Type 1.5 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Seattle Institute for Biomedical and Clinical Research (Other); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16707-D; 496539-188;; 16707D (Other: University of Washington)
Record Dates: First submitted 2005-09-14; First posted 2005-09-19 (Estimated); Results first posted 2011-08-10 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: type 2 diabetes mellitus; autoantibodies; islet proteins; rosiglitazone; glyburide; c-peptide
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Rosiglitazone; Glyburide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rosiglitazone (Active Comparator): Rosiglitazone is an oral antidiabetic agent which acts primarily by increasing insulin sensitivity. The rosiglitazone treatment group commenced therapy with 4 mg once per day and increase to twice per day if adequate glycemic control was not achieved.
  Interventions: Drug: rosiglitazone
- glyburide (Active Comparator): Glyburide is a sulfonylurea. Glyburide therapy was initiated with 2.5 mg in the morning or the patient was maintained on the dose they had been receiving prior to starting the study. This starting dose was raised by 2.5 in the evening and further up to a maximum of 10 mg twice a day if necessary to achieve desired glycemic control.
  Interventions: Drug: glyburide

INTERVENTIONS:
Drug: rosiglitazone — Tablet taken orally at a dosage of 4 mg once per day and increase to twice per day if adequate glycemic control was not achieved. Study drug was taken up to 3 years.
  Other Names: Avandia
  Arms: rosiglitazone
Drug: glyburide — Tablet taken orally, initially 2.5 mg in the morning or dose subject received prior to starting the study. Dosage was increased by 2.5 mg in the evening up to a maximum of 10 mg twice a day if necessary to achieve desired glycemic control. Study drug was taken up to 3 years.
  Arms: glyburide

SUMMARY:
The purpose of this research was to test whether one treatment was superior over another in the management of type 1.5 diabetes. Specifically we tested recently diagnosed antibody positive type 2 diabetic patients to determine whether treatment with rosiglitazone results in greater preservation of beta cell function compared to treatment with glyburide.

DETAILED DESCRIPTION:
Type 1 diabetes and Type 2 diabetes have different underlying pathophysiologic processes. The disease process in classical Type 1 diabetes is an autoimmune destruction of the pancreatic beta cells. In contrast, the disease process in classical Type 2 diabetes is not autoimmune in nature, a decreased sensitivity to insulin action is central to the disease process, and a poorly understood but non-inflammatory beta cell lesion occurs which diminishes insulin secretion. In clinical practice, the diagnosis of Type 1 versus Type 2 diabetes is made phenotypically using variables such as age at onset, apparent abruptness of onset of hyperglycemia, presence of ketosis, degree of obesity (especially central and intra abdominal), prevalence of other autoimmune diseases, and apparent need for insulin replacement. This clinical distinction of Type 1 versus Type 2 diabetes is recognized to be imperfect.

There is also a third group of individuals, who phenotypically are usually like classic Type 2 diabetics but who are positive for one or more of the autoantibodies commonly seen in the Type 1 disease process, namely islet cell antibodies (ICA) and/or insulin autoantibodies (IAA) and/or autoantibodies to glutamic acid decarboxylase (GAD Ab) and/or autoantibodies to the tyrosine phosphatase islet cell autoantibody 512 (IA 2 Ab).

These patients, autoantibody positive [Ab(+)] Type 2 or Type 1.5 diabetes, were the focus of our study. Compared to antibody negative Type 2 diabetics, patients with Type 1.5 diabetes have a more rapid decline in beta cell function, fail sulfonylurea therapy and require insulin therapy earlier (4-13).

Hypothesis: Rosiglitazone treatment will ameliorate or slow the underlying disease process in antibody positive Type 2 diabetes.

Patients meeting the inclusion criteria came in for a baseline visit. The nature of the study was explained and informed consent obtained. A fasting blood sample was obtained for autoantibodies, glucose, C peptide of proinsulin molecule (C-peptide), glycosylated hemoglobin (HbA1c), genetic typing, and T lymphocyte (T cell) responses to islet antigens. The beta cell function test was performed. Patients were then randomized to either rosiglitazone or glyburide.

All patients were encouraged to perform self blood glucose monitoring twice per day, before breakfast and before dinner. The treatment goals for all patients was the same: before breakfast and before dinner blood sugar levels between 90-130 milligrams per deciliter (mg/dI) and HbA1c of less then 7% without severe hypoglycemia. Patients unable to reach goal with monotherapy had metformin (initially) or acarbose (secondarily) added, as there is no evidence to suggest that either affect beta-cell function.

The rosiglitazone treatment group commenced therapy with 4 milligram (mg) once per day and increased to twice per day if adequate glycemic control was not achieved. For glyburide, therapy was initiated with 2.5 mg in the morning or the patient was maintained on the dose they had been receiving prior to starting the study. The starting dose was raised by 2.5 mg in the evening and further up to a maximum of 10 mg twice a day if necessary to achieve desired glycemic control.

If adequate control, HbA1c less than 7%, was not achieved on glyburide or rosiglitazone monotherapy, metformin was added and the dose gradually increased as needed and tolerated to a maximum of 1000 mg twice daily. If necessary, acarbose was also used up to a maximum dose of 100 mg thrice daily as needed and tolerated.

After initiation of the study, patients were seen at 1 month and then every 3 months for up to 3 years. Those patients randomized to rosiglitazone had the liver enzyme alanine transaminase (ALT) monitored every 2 months. In addition, telephone contact was utilized to achieve and maintain glycemic goals. Each participant was followed for up to 3 years. Drs. Chiu and Palmer coordinated the study. If the patient and his/her private physician prefer, the treatment protocol was implemented by the patient's private physician.

ELIGIBILITY:
Inclusion Criteria:

* Age at onset of diabetes - 35-69 years old.
* No history of ketonuria or ketoacidosis.
* Not requiring insulin to achieve glycemic control.
* Not receiving more than two oral hypoglycemic agents.
* Not taking a thiazolidinedione agent.
* HbA1c in established patients (on an oral hypoglycemia agent for over 4 months) of greater than 6% and under 10%.
* Fasting c-peptide greater than or equal to 0.8 ng/ml.
* Women must be either post-menopausal or on adequate birth control (i.e. oral contraceptives, tubal ligation, hysterectomy, condoms, or diaphragm) or use abstinence.

Exclusion Criteria:

* Patients with history of chronic pancreatitis or other secondary causes of diabetes.
* Patients receiving systemic corticosteroids.
* Patients with severe systemic illness (e.g. recent MI, CHF or cerebral vascular disease).
* Creatinine greater than 1.4 or liver enzymes greater than 2 times the upper limits of normal.
* Not able to adhere to the protocol.

Ages: 35 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2000-02; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry P Palmer, MD, Principal Investigator — Seattle Institute for Biomedical & Clinical Research, University of Washington, DVA Puget Sound Health Care System
Locations (1):
- DVA Puget Sound Health Care System, Seattle, Washington, United States

REFERENCES:
- [Background] Lampeter EF, Homberg M, Quabeck K, Schaefer UW, Wernet P, Bertrams J, Grosse-Wilde H, Gries FA, Kolb H. Transfer of insulin-dependent diabetes between HLA-identical siblings by bone marrow transplantation. Lancet. 1993 May 15;341(8855):1243-4. doi: 10.1016/0140-6736(93)91148-f. PMID 8098394
- [Background] DeFronzo RA. Pathogenesis of type 2 (non-insulin dependent) diabetes mellitus: a balanced overview. Diabetologia. 1992 Apr;35(4):389-97. doi: 10.1007/BF00401208. No abstract available. PMID 1516769
- [Background] Porte D Jr. Banting lecture 1990. Beta-cells in type II diabetes mellitus. Diabetes. 1991 Feb;40(2):166-80. doi: 10.2337/diab.40.2.166. PMID 1991568
- [Background] Zimmet PZ, Tuomi T, Mackay IR, Rowley MJ, Knowles W, Cohen M, Lang DA. Latent autoimmune diabetes mellitus in adults (LADA): the role of antibodies to glutamic acid decarboxylase in diagnosis and prediction of insulin dependency. Diabet Med. 1994 Apr;11(3):299-303. doi: 10.1111/j.1464-5491.1994.tb00275.x. PMID 8033530
- [Background] Tuomi T, Groop LC, Zimmet PZ, Rowley MJ, Knowles W, Mackay IR. Antibodies to glutamic acid decarboxylase reveal latent autoimmune diabetes mellitus in adults with a non-insulin-dependent onset of disease. Diabetes. 1993 Feb;42(2):359-62. doi: 10.2337/diab.42.2.359. PMID 8425674
- [Background] Zimmet PZ. The pathogenesis and prevention of diabetes in adults. Genes, autoimmunity, and demography. Diabetes Care. 1995 Jul;18(7):1050-64. doi: 10.2337/diacare.18.7.1050. No abstract available. PMID 7555542
- [Background] Groop LC, Bottazzo GF, Doniach D. Islet cell antibodies identify latent type I diabetes in patients aged 35-75 years at diagnosis. Diabetes. 1986 Feb;35(2):237-41. doi: 10.2337/diab.35.2.237. PMID 3510930
- [Background] Groop L, Miettinen A, Groop PH, Meri S, Koskimies S, Bottazzo GF. Organ-specific autoimmunity and HLA-DR antigens as markers for beta-cell destruction in patients with type II diabetes. Diabetes. 1988 Jan;37(1):99-103. doi: 10.2337/diab.37.1.99. PMID 3275559
- [Background] Kobayashi T, Tamemoto K, Nakanishi K, Kato N, Okubo M, Kajio H, Sugimoto T, Murase T, Kosaka K. Immunogenetic and clinical characterization of slowly progressive IDDM. Diabetes Care. 1993 May;16(5):780-8. doi: 10.2337/diacare.16.5.780. PMID 8098691
- [Background] Kobayashi T. Subtype of insulin-dependent diabetes mellitus (IDDM) in Japan: slowly progressive IDDM--the clinical characteristics and pathogenesis of the syndrome. Diabetes Res Clin Pract. 1994 Oct;24 Suppl:S95-9. doi: 10.1016/0168-8227(94)90234-8. PMID 7859641
- [Background] Kobayashi T, Nakanishi K, Sugimoto T, Itoh T, Murase T, Kosaka K, Tsuji K. Maleness as risk factor for slowly progressive IDDM. Diabetes Care. 1989 Jan;12(1):7-11. doi: 10.2337/diacare.12.1.7. PMID 2653752
- [Background] Kobayashi T, Itoh T, Kosaka K, Sato K, Tsuji K. Time course of islet cell antibodies and beta-cell function in non-insulin-dependent stage of type I diabetes. Diabetes. 1987 Apr;36(4):510-7. doi: 10.2337/diab.36.4.510. PMID 3545950
- [Background] Nakanishi K, Kobayashi T, Sugimoto T, Murase T, Itoh T, Kosaka K. Predictive value of insulin autoantibodies for further progression of beta cell dysfunction in non-insulin-dependent diabetics. Diabetes Res. 1988 Nov;9(3):105-9. PMID 3072143
- [Background] Hao W, Li L, Mehta V, Lernmark A, Palmer JP. Functional state of the beta cell affects expression of both forms of glutamic acid decarboxylase. Pancreas. 1994 Sep;9(5):558-62. doi: 10.1097/00006676-199409000-00003. PMID 7809009
- [Background] Mehta V, Hao W, Brooks-Worrell BM, Palmer JP. The functional state of the beta cell modulates IL-1 and TNF-induced cytotoxicity. Lymphokine Cytokine Res. 1993 Aug;12(4):255-9. PMID 8218598
- [Background] Gotfredsen CF, Buschard K, Frandsen EK. Reduction of diabetes incidence of BB Wistar rats by early prophylactic insulin treatment of diabetes-prone animals. Diabetologia. 1985 Dec;28(12):933-5. doi: 10.1007/BF00703140. PMID 4092862
- [Background] Atkinson MA, Maclaren NK, Luchetta R. Insulitis and diabetes in NOD mice reduced by prophylactic insulin therapy. Diabetes. 1990 Aug;39(8):933-7. doi: 10.2337/diab.39.8.933. PMID 2197139
- [Background] Keller RJ, Eisenbarth GS, Jackson RA. Insulin prophylaxis in individuals at high risk of type I diabetes. Lancet. 1993 Apr 10;341(8850):927-8. doi: 10.1016/0140-6736(93)91215-8. PMID 8096268
- [Background] Effect of intensive therapy on residual beta-cell function in patients with type 1 diabetes in the diabetes control and complications trial. A randomized, controlled trial. The Diabetes Control and Complications Trial Research Group. Ann Intern Med. 1998 Apr 1;128(7):517-23. doi: 10.7326/0003-4819-128-7-199804010-00001. PMID 9518395
- [Background] Diabetes Prevention Trial--Type 1 Diabetes Study Group. Effects of insulin in relatives of patients with type 1 diabetes mellitus. N Engl J Med. 2002 May 30;346(22):1685-91. doi: 10.1056/NEJMoa012350. PMID 12037147
- [Background] Kobayashi T, Nakanishi K, Murase T, Kosaka K. Small doses of subcutaneous insulin as a strategy for preventing slowly progressive beta-cell failure in islet cell antibody-positive patients with clinical features of NIDDM. Diabetes. 1996 May;45(5):622-6. doi: 10.2337/diab.45.5.622. PMID 8621013
- [Background] Kobayashi T, Maruyama T, Shimada A, Kasuga A, Kanatsuka A, Takei I, Tanaka S, Yokoyama J. Insulin intervention to preserve beta cells in slowly progressive insulin-dependent (type 1) diabetes mellitus. Ann N Y Acad Sci. 2002 Apr;958:117-30. doi: 10.1111/j.1749-6632.2002.tb02954.x. PMID 12021091
- [Background] Kumar S, Boulton AJ, Beck-Nielsen H, Berthezene F, Muggeo M, Persson B, Spinas GA, Donoghue S, Lettis S, Stewart-Long P. Troglitazone, an insulin action enhancer, improves metabolic control in NIDDM patients. Troglitazone Study Group. Diabetologia. 1996 Jun;39(6):701-9. doi: 10.1007/BF00418542. PMID 8781766
- [Background] Antonucci T, Whitcomb R, McLain R, Lockwood D, Norris RM. Impaired glucose tolerance is normalized by treatment with the thiazolidinedione troglitazone. Diabetes Care. 1997 Feb;20(2):188-93. doi: 10.2337/diacare.20.2.188. PMID 9118772
- [Background] Nolan JJ, Ludvik B, Beerdsen P, Joyce M, Olefsky J. Improvement in glucose tolerance and insulin resistance in obese subjects treated with troglitazone. N Engl J Med. 1994 Nov 3;331(18):1188-93. doi: 10.1056/NEJM199411033311803. PMID 7935656
- [Background] Nakanishi K, Kobayashi T, Miyashita H, Ohkubo M, Sugimoto T, Murase T, Kosaka K, Inouye K, Kono M. Relationships among islet cell antibodies, residual beta-cell function, and metabolic control in patients with insulin-dependent diabetes mellitus of long duration: use of a sensitive C-peptide radioimmunoassay. Metabolism. 1990 Sep;39(9):925-30. doi: 10.1016/0026-0495(90)90302-s. PMID 2202883
- [Background] Nakanishi K, Kobayashi T, Inoko H, Tsuji K, Murase T, Kosaka K. Residual beta-cell function and HLA-A24 in IDDM. Markers of glycemic control and subsequent development of diabetic retinopathy. Diabetes. 1995 Nov;44(11):1334-9. doi: 10.2337/diab.44.11.1334. PMID 7589833
- [Background] Sjoberg S, Gunnarsson R, Gjotterberg M, Lefvert AK, Persson A, Ostman J. Residual insulin production, glycaemic control and prevalence of microvascular lesions and polyneuropathy in long-term type 1 (insulin-dependent) diabetes mellitus. Diabetologia. 1987 Apr;30(4):208-13. doi: 10.1007/BF00270417. PMID 3297896
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] Juneja R, Hirsch IB, Naik RG, Brooks-Worrell BM, Greenbaum CJ, Palmer JP. Islet cell antibodies and glutamic acid decarboxylase antibodies, but not the clinical phenotype, help to identify type 1(1/2) diabetes in patients presenting with type 2 diabetes. Metabolism. 2001 Sep;50(9):1008-13. doi: 10.1053/meta.2001.25654. PMID 11555830
- [Background] Brooks-Worrell BM, Juneja R, Minokadeh A, Greenbaum CJ, Palmer JP. Cellular immune responses to human islet proteins in antibody-positive type 2 diabetic patients. Diabetes. 1999 May;48(5):983-8. doi: 10.2337/diabetes.48.5.983. PMID 10331401
- [Background] Gleichmann H, Zorcher B, Greulich B, Gries FA, Henrichs HR, Betrams J, Kolb H. Correlation of islet cell antibodies and HLA-DR phenotypes with diabetes mellitus in adults. Diabetologia. 1984 Jul;27 Suppl:90-2. doi: 10.1007/BF00275656. PMID 6383926
- [Background] Hagopian WA, Karlsen AE, Gottsater A, Landin-Olsson M, Grubin CE, Sundkvist G, Petersen JS, Boel E, Dyrberg T, Lernmark A. Quantitative assay using recombinant human islet glutamic acid decarboxylase (GAD65) shows that 64K autoantibody positivity at onset predicts diabetes type. J Clin Invest. 1993 Jan;91(1):368-74. doi: 10.1172/JCI116195. PMID 8423232
- [Background] Rowley MJ, Mackay IR, Chen QY, Knowles WJ, Zimmet PZ. Antibodies to glutamic acid decarboxylase discriminate major types of diabetes mellitus. Diabetes. 1992 Apr;41(4):548-51. doi: 10.2337/diab.41.4.548. PMID 1607079
- [Derived] Brooks-Worrell BM, Palmer JP. Attenuation of islet-specific T cell responses is associated with C-peptide improvement in autoimmune type 2 diabetes patients. Clin Exp Immunol. 2013 Feb;171(2):164-70. doi: 10.1111/cei.12012. PMID 23286943

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited through endocrinology physicians.
Groups:
- Rosiglitazone Autoantibody Positive: Rosiglitazone is an oral antidiabetic agent which acts primarily by increasing insulin sensitivity. The rosiglitazone treatment group commenced therapy with 4 milligram (mg) once per day and increase to twice per day if adequate glycemic control was not achieved. Autoantibody positive for one or multiple islet autoantibodies. These autoantibodies include insulin autoantibodies(IAA), islet cell autoantibodies (ICA), glutamic acid decarboxylase (GAD),and/or islet cell autoantibodies 512 (IA2).
- Rosiglitazone Autoantibody Negative: Rosiglitazone is an oral antidiabetic agent which acts primarily by increasing insulin sensitivity. The rosiglitazone treatment group commenced therapy with 4 mg once per day and increase to twice per day if adequate glycemic control was not achieved. Autoantibody negative for insulin autoantibodies (IAA), islet cell autoantibodies (ICA), glutamic acid decarboxylase (GAD), and islet cell autoantibodies 512 (IA2).
- Glyburide Autoantibody Positive: Glyburide is a sulfonylurea. Glyburide therapy was initiated with 2.5 mg in the morning or the patient was maintained on the dose they had been receiving prior to starting the study. This starting dose was raised by 2.5 in the evening and further up to a maximum of 10 mg twice a day if necessary to achieve desired glycemic control. Autoantibody positive for one or multiple islet autoantibodies. These autoantibodies include insulin autoantibodies(IAA), islet cell autoantibodies (ICA), glutamic acid decarboxylase (GAD), islet cell autoantibodies 512 (IA2).
- Glyburide Autoantibody Negative: Glyburide is a sulfonylurea. Glyburide therapy was initiated with 2.5 mg in the morning or the patient was maintained on the dose they had been receiving prior to starting the study. This starting dose was raised by 2.5 in the evening and further up to a maximum of 10 mg twice a day if necessary to achieve desired glycemic control. Autoantibody negative for insulin autoantibodies (IAA), islet cell autoantibodies (ICA), glutamic acid decarboxylase (GAD), and islet cell autoantibodies 512 (IA2).
Period: Overall Study
Arm/Group | Rosiglitazone Autoantibody Positive | Rosiglitazone Autoantibody Negative | Glyburide Autoantibody Positive | Glyburide Autoantibody Negative
Started | 15 | 15 | 13 | 21
Completed | 4 | 10 | 7 | 9
Not Completed | 11 | 5 | 6 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rosiglitazone Autoantibody Positive | Rosiglitazone Autoantibody Negative | Glyburide Autoantibody Positive | Glyburide Autoantibody Negative | Total
Number analyzed (Participants) | 15 | 15 | 13 | 21 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 13 | 12 | 18 | 57
  >=65 years | 1 | 2 | 1 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (8.8) | 56.4 (8.7) | 53.7 (9) | 57.5 (6.9) | 55.8 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 2 | 8 | 18
  Male | 11 | 11 | 11 | 13 | 46
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 13 | 21 | 64

OUTCOME MEASURES:

1. Primary Outcome: Changes in Beta Cell Function Assessed by Fasting and Stimulated C-peptide Measured at 36 Months.
Description: Changes in beta cell function assessed by fasting and stimulated C-peptide measured at 36 months.
Time Frame: 36 months
Population: Analysis per protocol
Measure: Mean (Standard Deviation); unit: ng per ml
Arm/Group | Rosiglitazone Autoantibody Positive | Rosiglitazone Autoantibody Negative | Glyburide Autoantibody Positive | Glyburide Autoantibody Negative
Number analyzed (Participants) | 15 | 15 | 13 | 21
ng per ml
  Fasting C-peptide | -0.4 (1.0) | -1.4 (1.6) | 0.1 (1.2) | 0.3 (1.1)
  Glucagon Stimulated C-peptide | -0.6 (1.6) | -2.8 (2.5) | 3.1 (12.1) | 0.3 (2.2)

2. Secondary Outcome: Patients Positive for T Cell Responses to Islet Proteins at 36 Months.
Description: Number of participants positive for T cell reactivity to islet proteins at 36 months.
Time Frame: 36 months
Measure: Number; unit: participants
Arm/Group | Rosiglitazone Autoantibody Positive | Rosiglitazone Autoantibody Negative | Glyburide Autoantibody Positive | Glyburide Autoantibody Negative
Number analyzed (Participants) | 4 | 10 | 7 | 9
participants | 1 (0) | 2 (0) | 2 (0) | 3 (0)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the period the research subjects were actively participating in the study. This time period was between February 3, 2000 through September 8, 2008.
Arm/Group | Rosiglitazone Autoantibody Positive | Rosiglitazone Autoantibody Negative | Glyburide Autoantibody Positive | Glyburide Autoantibody Negative
Serious Adverse Events (participants affected / at risk) | 1/15 | 2/15 | 0/13 | 3/21
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 1/13 | 1/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rosiglitazone Autoantibody Positive (N=15) | Rosiglitazone Autoantibody Negative (N=15) | Glyburide Autoantibody Positive (N=13) | Glyburide Autoantibody Negative (N=21)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Hypertension and diabetes related. Unknown if related to study.
Cholecystitis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unknown if study related.
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unknown if related to study.
Stroke (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Unknown if related to study.
Heart Attack (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Unknown if related to study.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rosiglitazone Autoantibody Positive (N=15) | Rosiglitazone Autoantibody Negative (N=15) | Glyburide Autoantibody Positive (N=13) | Glyburide Autoantibody Negative (N=21)
Hypoglycemia (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Small numbers based on high drop out of participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes